CLINICAL TRIAL: NCT05647161
Title: A Multicenter, Randomized, Controlled Study to Evaluate the Safety and Efficacy of the Adhesion Prevention Device BAX602 in Preventing the Adhesion Around Great Cardiac Vessels in Pediatric Patients With Congenital Heart Disease Undergoing Re-do Open Heart Surgery
Brief Title: BAX602 in Preventing the Adhesion Around Great Cardiac Vessels in Pediatric Patients With Congenital Heart Disease Undergoing Re-do Open Heart Surgery (Japan Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAX602-PED
Record Dates: First submitted 2022-11-18; First posted 2022-12-12 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Congenital Heart Disease in Children
Keywords: open heart surgery; anti-adhesion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Participants undergo 1st open heart surgery (first operation), and before closing the chest BAX602 will be sprayed on the surface of the heart and large vessels. Efficacy will be evaluated via adhesiolysis after re-do (2nd) open heart surgery.
  Re-do open (2nd) heart surgery will be performed ≥3 month (90 days) to ≤12 months (360 days) after 1st open heart surgery. If the re-do open heart surgery is performed later than 12 months (360 days) after the 1st open heart surgery, serious adverse events should be collected until the end of the clinical trial (at the time of discharge after re-do surgery), all observations and endpoints will be collected, including primary endpoints, items related to secondary endpoints, safety endpoints, and other observational items whenever possible. The participants will be observed for safety up to discharge after re-do open heart surgery (up to 30 days).
  Interventions: Device: BAX602
- Non-Treatment Group (Active Comparator): Participants undergo 1st open heart surgery (first operation) and the chest will be closed without spraying BAX602. Efficacy will be evaluated via adhesiolysis after re-do (2nd) open heart surgery.
  Re-do open (2nd) heart surgery will be performed ≥3 month (90 days) to ≤12 months (360 days) after 1st open heart surgery. If the re-do open heart surgery is performed later than 12 months (360 days) after the 1st open heart surgery, serious adverse events should be collected until the end of the clinical trial (at the time of discharge after re-do surgery), all observations and endpoints will be collected, including primary endpoints, items related to secondary endpoints, safety endpoints, and other observational items whenever possible. The participants will be observed for safety up to discharge after re-do open heart surgery (up to 30 days).
  Interventions: Device: No Intervention

INTERVENTIONS:
Device: BAX602 — Consists of the spray agent, spray set, and spraying device (regulator). Dissolves a polyethylene glycol (PEG) derivative with an N-hydroxysuccinimide group at the end (COH102) and a PEG derivative with a thiol group (COH206) as an anti-adhesion agent, which is sprayed on the surgical surface to reduce the degree, frequency, and extent of organ adhesions after surgery.
  Arms: Treatment Group
Device: No Intervention — Control Group
  Arms: Non-Treatment Group

SUMMARY:
Congenital heart disease occurs in about 1% of live births and can range from (1) naturally curable conditions that require no treatment to (2) conditions that require multiple immediate operations or refractory severe conditions. In the course of a staged surgical intervention, adhesion formation around the heart and large vessels can occur, and dissection of the adhesion site is required at the time of reoperation. There is a concern that dissection may markedly increase the risk of operation such as prolonged surgical time, cardiovascular injury, and increased blood loss, and medical devices to prevent adhesion formation after operation in the field of pediatric cardiovascular operation are strongly desired in medical settings.

The investigational product (BAX602), which has already been manufactured and marketed by Baxter overseas, has been used for open heart surgery as a local hemostatic agent without biological materials in Europe and the US for more than 20 years.

However, since it has not been approved in Japan, this randomized controlled study will be conducted in Japan to demonstrate the effect of BAX602 to prevent and reduce adhesion formation between the surface of the heart/large vessels and surrounding tissues in pediatric patients undergoing planned multistage operation for congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients <12 years of age
2. Patients who have undergone the first scheduled palliative surgery for the following diseases and are scheduled to undergo re-do open heart surgery (anatomical repair surgery):

   * Ventricular septal defect
   * Atrioventricular septal defect
   * Tetralogy of Fallot (spectrum)
   * Single ventricle disease (The participant should not meet the exclusion criteria (1) to (3)).
3. Patients who will undergo BT shunting or pulmonary artery banding (including bilateral pulmonary artery banding) for the first surgery
4. Patients undergoing repair surgery (anatomical repair surgery) or bi-directional Glenn surgery as the second target procedure
5. Patients for whom written consent has been obtained from the patient or a surrogate

Exclusion Criteria:

1. Patients with hypoplastic left heart syndrome (HLHS) and its analogues.
2. Patients with asplenia or hypersplenism.
3. Patients undergoing Norwood surgery as the second surgery.
4. Patients undergoing open heart surgery prior to the first scheduled palliative surgery.
5. Patients with complications of other organs that affect the indication for cardiac surgery.
6. Patients with chromosomal or genetic abnormalities that may affect the indication for cardiac surgery.
7. Patients with severe infections or multiple organ failure.
8. Patients who require emergency surgery that requires emergency life support.
9. Patients' body weight is less than 2,500g at birth.
10. Patients who are participating in other clinical trials or who are scheduled to participate in other clinical trials during this study period.
11. Patients who are judged by the investigator or sub investigator to be inappropriate to participate in this study for other reasons.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Grade of adhesion between the surface of the heart/large vessels and surrounding tissues | Day 90 to Day 360 (2nd open heart surgery)
  The following score of adhesion grade will be used:
  Grade 0=No adhesions; Grade 1=Filmy and avascular; Grade 3=Filmy, noncohesive requiring blunt and sharp dissection; Grade 4=Dense and cohesive requiring extensive sharp dissection.
  Lower score is better outcome.

SECONDARY OUTCOMES:
Total surgery time | Day 90 to Day 360 (2nd open heart surgery)
Time from start of skin incision to start of extracorporeal circulation | Day 90 to Day 360 (2nd open heart surgery)
Time from start of skin incision to the end of adhesion dissection | Day 90 to Day 360 (2nd open heart surgery)
Total score of grade of adhesion at evaluation sites | Day 90 to Day 360 (2nd open heart surgery)
  The following score of adhesion grade will be used:
  Grade 0=No adhesions; Grade 1=Filmy and avascular; Grade 3=Filmy, noncohesive requiring blunt and sharp dissection; Grade 4=Dense and cohesive requiring extensive sharp dissection.
  Lower score is better outcome.
  Adhesion will be evaluated at the following six sites.
  1. Pericardiotomy incision line area
  2. Anterior surface of the right ventricle
  3. Ascending aorta area
  4. Right atrial appendage
  5. Right atrial body
  6. Diaphragmatic surface
Grade of adhesion by evaluation site and presence or absence of extracorporeal circulation | Day 90 to Day 360 (2nd open heart surgery)
Number of sites of Grades ≥1, ≥2, ≥3, or 4 of adhesion | Day 90 to Day 360 (2nd open heart surgery)
Number of participants with sites of Grades ≥1, ≥2, ≥3, or 4 of adhesion | Day 90 to Day 360 (2nd open heart surgery)
Worst grade of adhesion by participants | Day 90 to Day 360 (2nd open heart surgery)
Intraoperative breeding amount | Day 90 to Day 360 (2nd open heart surgery)
Number of participants by type of local hemostatic agent used during surgery | Day 90 to Day 360 (2nd open heart surgery)

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Aichi Children's Hospital and Medical Center, Ōbu, Aichi-ken
  - Fukuoka Children's Hospital, Fukuoka, Fukuoka
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Nagano Children's Hospital, Azumino, Nagano
  - Okayama University Hospital, Okayama, Okayama-ken
  - Shizuoka Children's Hospital, Shizuoka, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: https://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy